CLINICAL TRIAL: NCT05388396
Title: Pediatric Inflammatory Multisystem Syndrome (PIMS-TS) in Pediatric Intensive Care: Retrospective Cohort Trial
Brief Title: PIMS-TS in Intensive Care: Retrospective Cohort Trial
Acronym: PIMS-TS INT
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: University Hospital, Motol (Other); Department of Anaesthesiology and Intensive CareMedicine, The Donaustadt Clinic, Lango Bardenstraße 122, 1220 Vienna, Austria (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: PIMS-TS INT
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Pims-Ts
Keywords: PIMS-TS; children; child; intensive care; critical illness
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PIMS-TS patients: Pediatric patients with PIMS-TS admitted to the PICU in selected time period
  Interventions: Other: PIMS-TS diagnostic a treatment

INTERVENTIONS:
Other: PIMS-TS diagnostic a treatment — PIMS-TS diagnostic a treatment

SUMMARY:
Pediatric Multisystem Inflammatory Syndrome Temporally associated with SARS-CoV-2, (PMIS-TS) represents the new unit, partially imitating the previously described Kawasaki disease. Due to variable and frequently incomplete clinical presentation together with variable disease severity, the real incidence in pediatric population remains unclear. Currently, PIMS-TS is defined by persistent fever, elevation of inflammatory markers, organ dysfunction (cardiac, central nervous system, respiratory, coagulation, renal, gastrointestinal), skin lesions (exanthematous), and absence of other possible etiology.

DETAILED DESCRIPTION:
During the world COVID-19 pandemic (2020-2022), pediatric patients with PIMS-TS represented a significant part of pediatric intensive care unit (PICU) load. The initial clinical presentation of patients with PIMS-TS could vary significantly, and also due to progressively evolving recommendations, the diagnostic a therapy could vary regionally and over the time too. The aim of this retrospective cohort trial was to describe the initial clinical presentation, diagnostics, therapy and clinical outcome of pediatric patients admitted during 2020-2022 to the one of the 3 university hospital PICUs.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with PIMS-TS
* PICU admission

Exclusion Criteria:

* insufficient data
* patients not admitted to PICU

Max Age: 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients with PIMS-TS admitted to PICU
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Initial clinical presentation | During the first 24 hours after PICU admission
  Vital signs
Initial laboratory results | During the first 24 hours after PICU admission
PIMS-TS treatment | During the first month after PICU admission
  PIMS-TS treatment specification

SECONDARY OUTCOMES:
PIMS-TS outcome | after one month from hospital discharge
  clinical and cardiology outcome after 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided